CLINICAL TRIAL: NCT05923632
Title: The Effect Of Model-Based Dıgıtal Game On Metabolıc Control, Self-Effıcıency And Qualıty Of Lıfe In Chıldren Wıth Type 1 Dıabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Bedriye AK, Assosiciate Prof. Dr., Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AİBÜ-HEM-BA-01
Record Dates: First submitted 2023-05-05; First posted 2023-06-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Children, Only
Keywords: Type 1 Diabetes; Children; Digital Game; Metabolic Control; Self-efficacy; Life Quality
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Who will be assigned to the experimental or control group will be determined by using the "https://www.randomizer.org/" site. Blinding will be done at the beginning of the research when assigning groups and in the statistics and reporting part. At the end of the study, measures will be taken to prevent bias in the measurement in the coding of the data and the evaluation of the statistician. The statistician will not be informed whether the groups are experiments or controls. To avoid bias in the evaluation of data; It is thought that the statistical analyzes of the coded data in the prepared database will be done by a statistics and operations expert independent of the researcher. Data entries will be entered with "A" and "B" codes without specifying the experimental or control group, and the analysis of the data will be done by coding as "A" and "B" groups. After the statistical analysis, the coding of the experimental and control groups will be explained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric patients with type 1 diabetes (Experimental): By providing standard diabetes education before the digital game intervention, the child who enters the game will be asked to fill out the Child with Type 1 Diabetes Descriptive Information Form, the Quality of Life in Children with Type 1 Diabetes Scale, and the Diabetes Management Self-Efficacy Scale in Children with Type 1 Diabetes.After the children in the experimental group are informed about the digital game designed according to the Information-Motivation-Behavioral Skills Model (IIMB) in diabetes management, active participation of the children in the digital game will be ensured for 9 weeks, and participation status will be followed in the background of the game.At the end of 9 weeks, children will be asked to complete all stages of the game.Children who do not complete the game will be contacted once a week in line with the follow-up, and reminders will be made.At the 12th and 15th weeks (3 and 6 weeks after the training), all the scales will be administered again.
  Interventions: Behavioral: Dijital Game and Health Education
- Pediatric patients with type 1 diabetes receiving routine care (No Intervention): At the beginning of the study, standard diabetes education will be given, and they will be asked to fill out the Children with Type 1 Diabetes Information Form, the Quality of Life Scale for Children with Type 1 Diabetes, and the Diabetes Management Self-Efficacy Scale. All scales will be administered again in the 12th and 15th weeks from the beginning of the study.

INTERVENTIONS:
Behavioral: Dijital Game and Health Education — After the children in the experimental group are informed about the digital game designed according to The The Information-Motivation-Behavioral Skills Model (IMB) in diabetes management, active participation of the children in the digital game will be ensured for 9 weeks; and participation status will be followed in the background of the game. At the end of 9 weeks, children will be asked to complete all stages of the game. Children who do not complete the game will be contacted once a week in line with their background follow-up and reminders will be made.
  Arms: Pediatric patients with type 1 diabetes

SUMMARY:
This study was planned to determine the effect of model-based digital game on metabolic control, self-efficacy and quality of life in children with T1DM.

DETAILED DESCRIPTION:
This study was planned to determine the effect of model-based digital game on metabolic control, self-efficacy and quality of life in children with T1DM. This study was planned as a randomized controlled trial with a pre-post test parallel group. Participants to be included in the study, In this study, children between the ages of 8-13 who were diagnosed with T1DM and followed up in the Pediatric Endocrinology outpatient clinics and services of two hospitals in two different centers will be selected. During the follow-up days of the children in the outpatient clinic, the diabetes nurse will be contacted to discuss working with the child with T1DM and their families. After the child and their parents are informed about the purpose and application of the study, that the collected data will only be used for scientific research purposes, the children and their families who gave their consent to participate in the study will be asked to sign the volunteering form. Children who agree to participate in the study will be given a password to log in to the created web page. Experimental and control groups will be determined according to the order of login with this password and randomization with https://www.randomizer.org/. Standard diabetes education was given to both groups before the game intervention to be applied to the experimental group; Children entering the site will be asked to fill in the Child with Type 1 Diabetes Descriptive Information Form, the Quality of Life in Children with Type 1 Diabetes Scale and the Diabetes Management Self-Efficacy Scale in Children with Type 1 Diabetes. After informing the children in the experimental group about the game designed based on The Information-Motivation-Behavioral Skills Model(IMB) of diabetes management on the website, it will be ensured that the children actively participate in the game for 9 weeks and their participation status in the background of the game will be followed; At the end of 9 weeks, all stages of the game will be required to be completed. Reminders will be made by contacting the children who have not completed the game in line with the follow-ups in the background, once a week. During this process, the control group; On a weekly basis, slides supported with visuals related to nutrition, exercise and drug use will be presented on the web page in the form of sessions. Children will be provided to watch each session. Whether the children complete the sessions or not will be monitored from the background. Children who do not complete the sessions will be reminded once a week.

All scales will be re-administered to both groups at the 12th week (3 weeks after the training). Scales will also be applied through the website. HbA1c and other blood levels of the parameters to be used in the study will be obtained from the hospital files at the beginning of the study and at the end of the 12th week, as they are routinely requested during the controls. At the end of the study, the control group will also be allowed to log in to the game via the website in terms of ethical compliance.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 8-13 age range,
* Being diagnosed with T1DM at least 6 months ago,
* Ability to read and write Turkish,
* Ability to communicate verbally,
* To have Internet access,
* Computer, tablet, etc. to have and use technological tools,
* To volunteer to participate in the study

Exclusion Criteria:

• Having another chronic disease other than T1DM

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale for Children with Type 1 Diabetes (PedsQL 3.0) | 30 minutes
  The scale was developed by Varni et al in 2003. It consists of five sub-dimensions: diabetes symptoms, treatment barriers, adherence to treatment, anxiety, and communication. The scale was prepared in a five-point Likert type, and the child form of the scale was designed for 5-7 age groups, 8-12 age groups and 13-18 age groups. A high total score from the scale indicates a high health-related quality of life. The internal consistency coefficient of the original form of the scale was 0.71(Varni et al,2003). The Turkish validity and reliability study of the 8-12 age form of the scale was performed by Ayar(2012), and the Turkish validity and reliability study of the 13-18 age form was performed by Çövener Özçelik et al(2015). In the study, the Cronbach's alpha values of the scales were 0.83 for 8-12 years old, 0.90 for 13-18 years old. In the studies of Ayar and Öztürk(2016); The internal consistency coefficient of the quality of life scale in children with diabetes was found to be 0.80.

SECONDARY OUTCOMES:
Diabetes Management Self-Efficacy Scale in Adolescents with Type 1 Diabetes | 30 minutes
  It is a scale developed by Moens(1998). In the scale prepared according to the fivepoint Likert system, 1= yes definitely, 2= maybe yes, 3=maybe yes, maybe no, 4=maybe no, 5 = of course no. The perceived self-efficacy score is calculated by dividing the total number of items, and there is a negative correlation between the increase in the total score and the level of self-efficacy. Medical treatment and nutrition (1-2-4-5-7-9-10-11-14-18-22-26); adjustment of nutrition and insulin dose (6-8-12-13-17-19-21-25); being able to tell about diabetes (23-24); it consists of four sub-dimensions, being honest with oneself and others(3-15-16-20). The total explanatory variance rate of the four-factor scale is 47.1%. The reliability coefficient of the original scale; It is 0.8.The Turkish validity and reliability study was done by Öztürk, Ayar and Bektas(2016). The total Cronbach's alpha coefficient of the Turkish scale is 0.85, and its sub-dimensions are 0.80, 0.75, 0.70 and 0.70, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Bedriye AK, Associate Prof.Dr., Study Director — Bolu Abant İzzet Baysal University; Özgür Bahadır, Lecturer, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (2):
- Turkey (Türkiye) (2):
  - Bolu Abant İzzet Baysal Üniversitesi, Bolu
  - Zonguldak Bülent Ecevit Üniversitesi, Zonguldak

IPD SHARING:
Plan to Share IPD: Yes
We wıll prepare the study as a thesıs. Then we wıll turn ıt ınto a publıcatıon ın an ınternatıonal magazıne.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data wıll be collected for 4 month
Access Criteria: Can be contacted through YOK-thesıs center

REFERENCES:
- [Background] Varni JW, Burwinkle TM, Jacobs JR, Gottschalk M, Kaufman F, Jones KL. The PedsQL in type 1 and type 2 diabetes: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales and type 1 Diabetes Module. Diabetes Care. 2003 Mar;26(3):631-7. doi: 10.2337/diacare.26.3.631. PMID 12610013
- [Background] Nansel TR, Weisberg-Benchell J, Wysocki T, Laffel L, Anderson B; Steering Committee of the Family Management of Diabetes Study. Quality of life in children with Type 1 diabetes: a comparison of general and diabetes-specific measures and support for a unitary diabetes quality-of-life construct. Diabet Med. 2008 Nov;25(11):1316-23. doi: 10.1111/j.1464-5491.2008.02574.x. PMID 19046222
- [Background] Christie D, Thompson R, Sawtell M, Allen E, Cairns J, Smith F, Jamieson E, Hargreaves K, Ingold A, Brooks L, Wiggins M, Oliver S, Jones R, Elbourne D, Santos A, Wong IC, O'Neill S, Strange V, Hindmarsh P, Annan F, Viner R. Structured, intensive education maximising engagement, motivation and long-term change for children and young people with diabetes: a cluster randomised controlled trial with integral process and economic evaluation - the CASCADE study. Health Technol Assess. 2014 Mar;18(20):1-202. doi: 10.3310/hta18200. PMID 24690402
- [Background] Brown SJ, Lieberman DA, Germeny BA, Fan YC, Wilson DM, Pasta DJ. Educational video game for juvenile diabetes: results of a controlled trial. Med Inform (Lond). 1997 Jan-Mar;22(1):77-89. doi: 10.3109/14639239709089835. PMID 9183781
- [Background] Gao J, Wang J, Zhu Y, Yu J. Validation of an information-motivation-behavioral skills model of self-care among Chinese adults with type 2 diabetes. BMC Public Health. 2013 Feb 4;13:100. doi: 10.1186/1471-2458-13-100. PMID 23379324
- [Background] Goncalves S, Barros V, Rui Gomes A. Eating-Disordered Behaviour in Adolescents with Type 1 Diabetes. Can J Diabetes. 2016 Apr;40(2):152-7. doi: 10.1016/j.jcjd.2015.09.011. Epub 2016 Feb 10. PMID 26874893
- [Background] Goyal S, Nunn CA, Rotondi M, Couperthwaite AB, Reiser S, Simone A, Katzman DK, Cafazzo JA, Palmert MR. A Mobile App for the Self-Management of Type 1 Diabetes Among Adolescents: A Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 Jun 19;5(6):e82. doi: 10.2196/mhealth.7336. PMID 28630037
- [Background] Holtz BE, Murray KM, Hershey DD, Dunneback JK, Cotten SR, Holmstrom AJ, Vyas A, Kaiser MK, Wood MA. Developing a Patient-Centered mHealth App: A Tool for Adolescents With Type 1 Diabetes and Their Parents. JMIR Mhealth Uhealth. 2017 Apr 19;5(4):e53. doi: 10.2196/mhealth.6654. PMID 28428167
- [Background] Johnson D, Deterding S, Kuhn KA, Staneva A, Stoyanov S, Hides L. Gamification for health and wellbeing: A systematic review of the literature. Internet Interv. 2016 Nov 2;6:89-106. doi: 10.1016/j.invent.2016.10.002. eCollection 2016 Nov. PMID 30135818
- [Background] Martos-Cabrera MB, Membrive-Jimenez MJ, Suleiman-Martos N, Mota-Romero E, Canadas-De la Fuente GA, Gomez-Urquiza JL, Albendin-Garcia L. Games and Health Education for Diabetes Control: A Systematic Review with Meta-Analysis. Healthcare (Basel). 2020 Oct 14;8(4):399. doi: 10.3390/healthcare8040399. PMID 33066372
- [Background] Nelson LA, Wallston KA, Kripalani S, LeStourgeon LM, Williamson SE, Mayberry LS. Assessing barriers to diabetes medication adherence using the Information-Motivation-Behavioral skills model. Diabetes Res Clin Pract. 2018 Aug;142:374-384. doi: 10.1016/j.diabres.2018.05.046. Epub 2018 Jun 4. PMID 29879495